CLINICAL TRIAL: NCT00287092
Title: A Randomised, Controlled, Double-Blind Study of the Immunogenicity and Safety of PEDIACEL®, a Combined Diphtheria, Tetanus, Five Component Acellular Pertussis, Inactivated Poliomyelitis and Haemophilus Influenzae Type b Conjugate Vaccine (Adsorbed) Compared To Infanrix®-IPV+Hib When Both Vaccines Are Given to Infants Using a Three Dose Immunisation Schedule ("Nordic Schedule" 3-5-12 Months)
Brief Title: Comparison of Safety and Immunogenicity of Pediacel™ and Infanrix™ IPV+Hib (Penta) Given in a 3 Dose Schedule in Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A5I15
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Pertussis; Diphtheria; Tetanus; Poliomyelitis; Haemophilus Influenzae Type b
Keywords: Haemophilus influenzae type b;; Corynebacterium diphtheriae;; Clostridium tetani;; Bordetella pertussis;; poliovirus types 1, 2 and 3;; Vero cell;; Influenza;; Diphtheria
MeSH Terms: conditions — Whooping Cough; Diphtheria; Tetanus; Poliomyelitis; Haemophilus Infections; Influenza, Human | interventions — diphtheria-tetanus-five component acellular pertussis-inactivated poliomyelitis -Haemophilus influenzae type b conjugate vaccine; Diphtheria-Tetanus-acellular Pertussis Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Group 1 (Experimental): Participants will receive PEDIACEL vaccine
  Interventions: Biological: DT5aP-IPV-Hib 5-component Pertussis vaccine
- Group 2 (Active Comparator): Participants will receive Infanrix-IPV+Hib vaccines
  Interventions: Biological: Infanrix® -IPV+Hib

INTERVENTIONS:
Biological: DT5aP-IPV-Hib 5-component Pertussis vaccine — 0.5 mL, IM
  Other Names: Pediacel™
  Arms: Group 1
Biological: Infanrix® -IPV+Hib — 0.5 mL, IM
  Other Names: Infanrix®
  Arms: Group 2

SUMMARY:
Pediacel™ is currently licensed in the UK for use as a 3 dose regimen for the active immunisation of infants against Diphtheria, Tetanus, Pertussis, Poliomyelitis and invasive infections caused by Haemophilus influenzae type b. However there are currently no clinical data supporting the use of Pediacel™ using a 3, 5, and 12 months of age vaccination schedule. This study is designed to provide safety and immunogenicity data to support the use of Pediacel™ according to a 3, 5, and 12 months schedule.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 80 to 120 days inclusive on the day of inclusion.
* Born at full term of pregnancy (> 37 weeks)
* Informed consent form signed by the parent(s) or other legal representative according to local regulations
* Parent(s) or legal representative able to attend all scheduled visits and to understand and comply with the study procedures (able to read and write; access to a telephone).

Exclusion Criteria:

* Rectal temperature ≥ 38.0°C
* Moderate or severe acute illness with or without fever
* Participation in another clinical trial in the 4 weeks preceding the first trial vaccination
* Having received any DTaP, IPV, or Hib vaccines prior to study initiation or any vaccination in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Known history of diphtheria, tetanus, pertussis, H. influenzae type b infections, poliomyelitis
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as long-term systemic corticosteroids therapy
* Systemic hypersensitivity to any of the vaccine components (including neomycin, streptomycin, polymyxin B and formaldehyde)
* History of a life-threatening reaction (such as encephalopathy, Hypotonic Hyporesponsive Episode, severe fever, convulsions, etc.) to the trial vaccine or a vaccine containing the same substances
* Blood or blood-derived products (immunoglobulins) received in the past 4 weeks
* Vaccination planned in the 6 weeks following any trial vaccination
* Known HIV seropositivity
* Thrombocytopenia or a bleeding disorder contraindicating intramuscular vaccination
* History of seizures or progressive, evolving or unstable neurological condition
* Clinically significant findings on review of systems that might interfere with correct vaccination or which, in the opinion of the Investigator, would interfere with the evaluation of the vaccine or pose a health risk to the subject.

Ages: 80 Days to 120 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 807 (Actual)
Dates: Start 2006-02; Primary Completion 2007-05 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the immunogenicity of PEDIACEL® Vaccine. | 1 Month post-dose 3

SECONDARY OUTCOMES:
To provide information concerning the safety after administration of PEDIACEL® Vaccine | Entire study period

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (12):
- Finland (11):
  - Espoo
  - Helsinki
  - Jarvenpaa
  - Jyväskylä
  - Kotka
  - Lahti
  - Oulu
  - Pori
  - Tampere
  - Turku
  - Vantaa
- Östersund, Sweden

REFERENCES:
- [Derived] Vesikari T, Silfverdal SA, Boisnard F, Thomas S, Mwawasi G, Reynolds D. Randomized, controlled, multicenter study of the immunogenicity and safety of a fully liquid combination diphtheria-tetanus toxoid-five-component acellular pertussis (DTaP5), inactivated poliovirus (IPV), and haemophilus influenzae type b (Hib) vaccine compared with a DTaP3-IPV/Hib vaccine administered at 3, 5, and 12 months of age. Clin Vaccine Immunol. 2013 Oct;20(10):1647-53. doi: 10.1128/CVI.00414-13. Epub 2013 Aug 21. PMID 23966556
- See also: Related Info — http://www.sanofipasteur.com